CLINICAL TRIAL: NCT03496285
Title: Multimodal MRI Study of Accumbofrontal Tract in Anorexia Nervosa and Obessional Compulsive Disorder : Search for Structural and Functional Changes Between Orbito-frontal Cortex and Accumbens Nucleus Subdivisions
Brief Title: Accumbofrontal Tract Study in 2 Populations of Patients With Anorexia Nervosa and Obsessional Compulsive Disorder and Healthy Volunteer
Acronym: ACCUMBENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ACCUMBENS
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Accumbo Frontal Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Multimodal MRI with diffusion sequence for anorexia nervosa patient — Multimodal MRI with diffusion sequence, resting state, T2, T1 without gadolinium contrast
Radiation: Multimodal MRI with diffusion sequence for obsessional compulsive disorder patient — Multimodal MRI with diffusion sequence, resting state, T2, T1 without gadolinium contrast
Radiation: Multimodal MRI with diffusion sequence for healthy volunteer — Multimodal MRI with diffusion sequence, resting state, T2, T1 without gadolinium contrast

SUMMARY:
Restrictive anorexia nervosa and TOCs are psychiatric diseases which shares a common pathophysiological substrate We hypothesize that anorexia patients and patients with OCD have structural and functional changes in the accumbofrontal tract. The main objective of this study will be to compare the structure and the connectivity of this tract in MRI with diffusion sequences (DTI tractography) and resting-state, in 3 distinct populations of anorexic patients, patients with OCD and healthy patients. The role of the accumbo-frontal tract in the cortico-striato-hypothalamo-cortical circuit seems to be established. DTI tractography will allow the measurement of functional anisotropy (FA), a parameter that evaluates the diffusion of water molecules along the white matter fibers, and therefore the potential alteration of the studied tract. Resting state sequences will allow to estimate the BOLD signal and the functionality of the tract.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age between 18 and 65 years
* Subjects free to give their written consent

For anorexia nervosa :

* Patients meeting the diagnostic criteria for anorexia nervosa according to DSM5 (American Psychiatric Association): low weight (<85% of expected weight for age and height), fear of gaining weight or becoming fat, distortion of body image, and amenorrhea for more than 3 months
* Treatment with at least one antidepressant and one anxiolytic

For OCD :

* Patients meeting the diagnostic criteria of OCDs according to DSM5 (American Psychiatric Association) : presence of obsessions and / or compulsions, resulting in clinically significant suffering (loss of at least one hour per day) or impairment at the social, occupational level or in another important area of life. These symptoms are not due to the physiological effects of a substance or a general medical condition and cannot be better explained by the symptoms of another psychiatric disorder.
* Patients with homogeneous OCD in obsession and compulsion.
* Normal weight compared to expected weight for age and height
* Treatment with at least one antidepressant and one anxiolytic

ForHealthy volunteer

•Normal weight compared to expected weight for age and height

Exclusion Criteria:

* Male
* Age <18 years or> 65 years
* Pregnancy
* Absence of free and informed consent signature
* Current processing by rTMS
* Somatic intercurrent pathologies: neurological, cardiological, pneumological, renal, hepatic, endocrine, metabolic disorders ...
* Mental retardation (WAIS-IV QI <70)
* Primary Amenorrhea
* Absolute contraindication or relative to the realization of a magnetic resonance imaging without injection of contrast medium
* Old or intercurrent psychotic pathology

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Fractional Anisotropy (probabilistic tractography) | 20 minutes
  Evaluate the mean functional anisotropy value for fiber bundles connecting the orbito-frontal cortex and the nucleus accumbens

SECONDARY OUTCOMES:
BOLD Signal (resting state) | 20 minutes
  Evaluate the value of the BOLD-signal of the fiber bundles connecting the orbito-frontal cortex and the nucleus accumbens

CONTACTS AND LOCATIONS:
Locations (1):
- CH Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No